CLINICAL TRIAL: NCT03122925
Title: Measurement of the TCA Cycle Rate in the Dentate Nucleus in Friedreich's Ataxia
Brief Title: TCA Cycle in the Dentate in Friedreich's Ataxia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: RAD-2017-25500
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: Healthy subjects
  Interventions: Device: MR
- Friedreich's Ataxia: Diagnosed for Friedreich's Ataxia
  Interventions: Device: MR

INTERVENTIONS:
Device: MR — MR

SUMMARY:
OBJECTIVE: To measure the tricarboxylic acid (TCA) cycle rate in the dentate nucleus in a group of control subjects and subjects with Friedreich's Ataxia (FRDA).

HYPOTHESIS: The TCA cycle rate will be lower in FRDA subjects than in controls APPROACH: The investigators will infuse carbon-13 (13C) labeled glucose and measure the rate of 13C label incorporation from glucose to glutamate in the brain using in vivo magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
The investigators will measure the TCA cycle rate in the dentate nucleus in a group of FRDA patients and in a group of age-matched healthy controls using 13C MRS in vivo together with systemic i.v. infusion of 13C-labeled glucose.

The investigators aim to obtain adequate data in 16 subjects grouped as follows:

* n=4 pilot subjects (healthy subjects) for testing and optimization of the experimental setup.
* n=6 healthy controls
* n=6 FRDA patients

In other to reach this goal, the investigators plan to recruit up to 20 subjects, in case some subjects withdraw before completion of the MR scan, or in case the measured data are not adequate (e.g. technical problem with the scanner).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to consent for themselves
* considered healthy (controls) OR be diagnosed with FRDA.

Exclusion Criteria:

* All subjects:
* Participants who cannot have an MRI, as determined by the CMRR safety screening form (e.g. metal implant)
* Pregnancy
* Clautrophobia
* Diabetes
* Clinically significant cardiac disease

Control subjects:

- Neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls Friedreich's Ataxia diagnosis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
TCA cycle rate in the dentate nucleus | Baseline
  value between 0 to 2 micromol/g/min

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Gilles Henry, PhD, Principal Investigator — University of Minnesota
Locations (1):
- CMRR, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No